CLINICAL TRIAL: NCT01931319
Title: Prevention of Baclofen Withdrawal Syndrome: Dose Escalation Study of Intravenous Baclofen in Healthy Adult Volunteers
Brief Title: Dose Escalation Study of Intravenous Baclofen in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Paralyzed Veterans of America Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baclofen_Dose escalation
Record Dates: First submitted 2013-08-14; First posted 2013-08-29 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Safety and Pharmacokinetics of Intravenous Baclofen
Keywords: baclofen withdrawal; interruption; spasticity; pharmacokinetics; tolerability; intravenous
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous Baclofen (Experimental): Three single doses were evaluated using three cohorts (N=12 per cohort). Subjects received single doses of baclofen: 7.5, 11.5 or 15mg 10-minute intravenous infusion administered over 10 minutes by an infusion pump and 10, 15, or 20mg taken orally with a 48-hour washout phase between oral and intravenous arms of the study. Initially, 3 subjects received study drug at a given dose, after assessing the safety and tolerance of baclofen the additional 9 subjects received study drug.
  Interventions: Drug: Intravenous baclofen

INTERVENTIONS:
Drug: Intravenous baclofen

SUMMARY:
The objective of this study is to determine safety and characterize pharmacokinetics of higher doses of intravenous baclofen in healthy subjects.

Thirty-six healthy adults received a single dose of PO baclofen (10mg, 15mg or 20mg) and a 10-minute infusion of IV baclofen (7.5mg, 11.5mg or 15mg respectively) with a minimum 48-hour wash out period. Twelve subjects also received a 60-minute infusion of 15mg IV baclofen following an additional 48-hour wash out period.

The pharmacokinetic and tolerability information gained from this study will support the development of further studies to assess the use of IV baclofen to prevent or treat baclofen withdrawal syndrome.

DETAILED DESCRIPTION:
This randomized, open-label, dose escalation, crossover study was conducted at a contract clinical research facility. Three single doses were evaluated using three cohorts (N=12 per cohort). Study doses were as follows: cohort 1 - 7.5mg IV and 10mg PO, cohort 2 - 11.5mg IV and 15mg PO, and cohort 3 - 15mg IV and 20mg PO. The IV baclofen doses for this trial were based on a 75% bioavailability observed in a previous low dose study.16 The oral formulation of the study drug used in this trial was 10mg baclofen tablet (Teva Pharmaceutical Industries Ltd.) and is commercially available. The intravenous formulation was 2mg/mL solution manufactured by Aptuit LLC. for this study. IV infusions were administered over 10 minutes. In addition, cohort 3 received 15mg over a 60-minute infusion. There was a minimum 48-hour washout period between doses. Initially, 3 subjects received study drug at a given dose, after assessing the safety and tolerance of baclofen the additional 9 subjects received study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18-65.
2. Subjects are capable of giving informed consent.
3. Female subjects must be post-menopausal for at least 1 year, or surgically incapable of bearing children, or practicing at least one or more of the following methods of contraception for three months prior to, and during the study: hormonal, intrauterine device (IUD), or barrier method in combination with a spermicide.
4. Subject should be medication free, other than hormonal birth control, for 48 hours before through 24 hours after study drug administration. If the need for medication is identified during this time period, it will be discussed with and approved by the PI.

Exclusion Criteria:

1. Women who are pregnant.
2. Women who are breastfeeding.
3. Subject has a history of intolerance to IV administration of medication.
4. Subject has a known hypersensitivity to baclofen.
5. Subject has a significant history of cardiac, neurologic, psychiatric, oncologic, endocrine, metabolic, renal or hepatic disease
6. Subject has taken or used any investigational drug or device in the 30 days prior to screening.
7. Subject has taken either prescribed or over the counter medication for 48 hours prior to baclofen administration on either of the study days, other than hormonal birth control.
8. Subject reveals clinically significant abnormalities on screening laboratory tests.
9. Subject is a non-English speaker, such that ability to ascertain neurological status would require an interpreter.
10. Sleep deprivation (for example. working the night shift the evening prior to the study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety assessments | Upto 24 hours following drug administration
  Blood Pressure & Pulse: Recorded every 5 minutes immediately prior to, and during the IV infusion, then every 15 minutes for 1 hour, then every hour for 12 hours.
  Assessment of sedation / sleepiness: Subjects will be assessed by using the sleepiness scale prior to drug administration then every 30 minutes for four hours after drug administration.
  Ataxia and nystagmus: Measured using the following rating scale and definitions of ataxia and nystagmus.
  0=none, 1=mild, 2=severe
  Ataxia: For those who are ambulatory, this will be assessed by gait. Ratings will be:
  mild-unsteady with tandem gait testing, but able to perform without assistance severe-unable to perform gait testing without assistance. For non-ambulatory subjects, ataxia will be assessed by finger to nose and finger pursuit maneuvers.
  Nystagmus:
  mild-present on extreme gaze; severe-present on midline gaze

SECONDARY OUTCOMES:
Maximum Concentration(Cmax) | Upto 24 hours following drug administration
  Cmax: Cmax is the maximum baclofen concentration observed
AUC(0-inf) | Upto 24 hours after drug administration
  AUC(0-inf): Area under the plasma concentration-versus-time curve from time zero to infinity
Plasma Decay Half-life (T1/2) | Up to 24 hours after drug administration
  Plasma Decay Half-life(T1/2): Plasma decay half-life is the time measured for the plasma concentration to decrease by one half

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Kriel, MD, Principal Investigator — University of Minnesota; James C Cloyd, PharmD, Principal Investigator — University of Minnesota; Linda E Krach, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States